CLINICAL TRIAL: NCT06435611
Title: Adiposity, Cardiometabolic and Neurocognitive Health Among Ethnic Groups: a Feasibility and Pilot Study (ACNH Study)
Brief Title: Adiposity, Cardiometabolic and Neurocognitive Health Among Ethnic Groups: a Feasibility and Pilot Study
Acronym: ACNH
Status: Recruiting | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Principal Investigator, Georgios Dimitriadis, Endocrinologist Consultant and Obesity Physician, King's College Hospital NHS Trust
Other Study IDs: 329603
Record Dates: First submitted 2023-07-12; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Metabolic Disease; Obesity; Hepatic Steato-Fibrosis; Cardiovascular Diseases; Cognitive Impairment
Keywords: obesity; multi-ethnicity; cardiovascular diseases; hepatic steatosis; metabolic diseases
MeSH Terms: conditions — Metabolic Diseases; Obesity; Cardiovascular Diseases; Cognitive Dysfunction; Fatty Liver

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this pilot and feasibility study is to is to test the feasibility of conducting a cross-sectional study on adiposity and cardiometabolic and neurocognitive risk factors at Kings College Hospital NHS Foundation Trust (KCH).

The main aim is to assess and compare anthropometric measurements of adiposity (weight, Body Mass Index (BMI), Waist Circumference (WC), Waist-to-Hip ratio (WHR), Neck circumference (NC)), liver fat (hepatic steatosis and fibrosis), cardiometabolic risk factors (dyslipidemia, insulin resistance, hypertension) and neurocognitive risk factors among participants, according to their ethnic background.

Participants will come at KCH for one visit and will have their anthropometric measurements and cardio-metabolic profile assessed. They will also perform questionnaires on lifestyle, socio-economic status and neuro-cognitive health during their visit.

DETAILED DESCRIPTION:
The first objective of this study is to test the feasibility of conducting a cross-sectional study on adiposity and cardiometabolic and neurocognitive risk factors at Kings College Hospital NHS Foundation Trust.

The second objective is to assess and compare anthropometric measurements of adiposity (weight, Body Mass Index (BMI), Waist Circumference (WC), Waist-to-Hip ratio (WHR), Neck circumference (NC)), liver fat (hepatic steatosis and fibrosis), cardiometabolic risk factors (dyslipidemia, insulin resistance, hypertension) and neurocognitive risk factors among participants, according to their ethnic background.

The third objective is to test the feasibility of assessing cognitive function, in relation to adiposity, by using standardised tests measuring cognitive function (MMSE, MoCA or an adapted version) among ethnic groups of various education levels and literacy, lifestyle and from different cultures. Our objective is also to test the feasibility of using lifestyle questionnaires [Food Frequencies Questionnaires (FFQ) and International Physical Activity Questionnaires -(IPAQ-S)] in various ethnic groups with regard to geographic variation (urban, rural).

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥18 years old
* Body mass index (BMI) ≥ 30 kg/m2

Exclusion Criteria:

* Severe obesity (BMI > 50 kg/m2)
* Pregnancy (positive urine hCG) or a recent pregnancy (in the past 6 months)
* Known active chronic hepatic diseases
* Known diagnosis of human immunodeficiency virus
* Pre-established diagnosis of advanced renal failure (estimated Glomerular Filtration Rate (eGFR) <30 ml/min)
* Diagnosis of decompensated heart failure
* History of bariatric surgery
* Uncontrolled thyroid disease
* Current use of the following medication: steroids (oral or injections only), weight-loss medication including over-the-counter products, glucagon-like peptide 1 (GLP-1) agonists , Sodium-Glucose Transport Protein 2 (SGLT2) Inhibitors

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult male and female living with obesity (BMI ≥ 30 kg/m2 )
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Height | 1 minute
  Measured without shoes and reported in centimeters
Insulin resistance | 10 minutes
  random plasma glucose, glycated haemoglobin (HbA1c) using a blood test
Type 2 Diabetes | 10 minutes
  random plasma glucose, glycated haemoglobin (HbA1c) using a blood test
Hepatic steatosis, and stages of fibrosis | 10 minutes
  Assessed by a certified physician using transient elastography (TE) measurements using a Fibroscan (Model mini-430).
neurocognitive risk factors | 15 minutes
  Result below 25 on the Montreal Cognitive Assessment test (MoCA). No minimum results, normal is above or equal to 26. The lower the result is the more the participant is at risk of presenting any form of neuro-cognitive impairment.
Weight | 1 minute
  Measured using an automatic scale, without shoes. Reported in kilograms.
BMI | 30 seconds
  Will be calculated from weight and height results and will be presented in kg/m2.
Waist circumference | 1 minute
  Will be measured with a tape around the middle point halfway between the top of the hips and the bottom of the ribs, at expiration. Will be reported in centimeters.
Hip circumference | 1 minute
  Will be measure with a tape around the widest part of the hips. Will be reported in centimeters.
Dyslipidemia | 10 minutes
  Will be diagnosed from lipid levels reported in a blood test
Neck circumference | 1 minutes
  Will be measure with a tape around a point just below the larynx (Adam's Apple) and perpendicular to the long axis of the neck. The participant should look straight ahead during measurement, with shoulders down (not hunched). Round the neck measurement up to nearest ½ centimeters. Result will be reported in centimeters.
Waist-to-Hip ratio | 30 seconds
  Will be derived from waist circumference and hip circumference.
Waist-to-Height ratio | 30 seconds
  Will be derived from waist circumference and height.
Hypertension (estimated using blood pressure measurement) | 10minutes
  blood pressure will consist of 3 systolic blood pressure and diastolic blood pressure measurements

CONTACTS AND LOCATIONS:
Overall Officials: Georgios K. Dimitriadis, PhD, Principal Investigator — Kings College Hospital
Locations (2):
- United Kingdom (2):
  - King's College Hospital NHS Foundation Trust, London, United Kingdom of Great Britain and Northern Ireland
  - King's College Hospital NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared among different collaborative centers to compare outcomes among different ethnic groups from rural and urban environment of low- middle and high income countries.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1 year
Access Criteria: To have collected 10 participants (5 males and 5 females) as per protocol and have agreed on a specific data sharing agreement signed by all parties.